CLINICAL TRIAL: NCT02419612
Title: A 52-week International, Multicenter, Randomized, Double-Blind, Active-Controlled, Parallel Group, Phase 3bTrial With a Blinded 104-week Long -Term Extension Period to Evaluate the Efficacy and Safety of Saxagliptin Co-administered With Dapagliflozin in Combination With Metformin Compared to Glimepiride in Combination With Metformin ≥1500 mg in Adult Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Therapy Alone
Brief Title: A 52-week International, Multicenter Trial With a Long -Term Extension to Evaluate Saxagliptin With Dapagliflozin in Combination With Metformin Compared to Glimepiride in Combination With Metformin in Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CV181-365
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — saxagliptin; dapagliflozin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin 5 mg/ dapagliflozin 10mg or Placebo (Experimental): Saxagliptin 5 mg /dapagliflozin 10 mg Placebo once a day orally
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin; Other: Placebo
- Glimepiride or Placebo (Experimental): Glimepiride or placebo 1mg or 2mg or 3mg or 4mg or 6mg once a day orally
  Interventions: Drug: Glimepiride; Other: Placebo

INTERVENTIONS:
Drug: Saxagliptin
  Arms: Saxagliptin 5 mg/ dapagliflozin 10mg or Placebo
Drug: Dapagliflozin
  Arms: Saxagliptin 5 mg/ dapagliflozin 10mg or Placebo
Drug: Glimepiride
  Arms: Glimepiride or Placebo
Other: Placebo

SUMMARY:
This clincial trial is evaluating if the co-administration of saxagliptin and dapagliflozin, in addition to metformin, results in better glycemic control, as measured by HbA1c, over a treatment period of 52 weeks, compared to the addition of glimepiride to metformin in subjects with Type 2 Diabetes Mellitus who have inadequate glycemic control on Metformin Alone. We will compare the change from baseline in HbA1c achieved with saxagliptin, in co-administration with dapagliflozin, added to current background therapy with metformin compared to glimepiride added to current background therapy with metformin ≥1500 mg at Week 52.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects must be willing and able to give signed and dated written informed consent
* Patients with Type 2 diabetes mellitus (T2DM) with inadequate glycemic control
* Subjects should have been taking the same daily dose of metformin ≥ 1500 mg
* Fasting Plasma Glucose ≤ 270 mg/dL (≤15 mmol/L)
* Males and females, aged ≥18 years old at time of screening visit
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test
* WOCBP and males must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug

Exclusion Criteria:

* Clinical diagnosis of type I diabetes
* History of diabetic ketoacidosis
* Cardiovascular/vascular diseases within 3 months of the enrollment
* Renal disease
* Hepatic diseases
* History of, or currently, acute or chronic pancreatitis
* Hematological and oncological disease/conditions
* Patients who have contraindications to therapy being studied
* Patients on weight loss program(s)
* Replacement or chronic systemic corticosteroid therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (70):
- United States (20):
  - Research Site, Birmingham, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Huntington Park, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, Tarzana, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Edina, Minnesota
  - Research Site, Las Vegas, Nevada
  - Research Site, Greer, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
- Czechia (6):
  - Research Site, Cheb
  - Research Site, Hradec Králové
  - Research Site, Krnov
  - Research Site, Kroměříž
  - Research Site, Náchod
  - Research Site, Prague
- Germany (2):
  - Research Site, Dresden
  - Research Site, Leipzig
- Hungary (10):
  - Research Site, Ajka
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
  - Research Site, Zalaegerszeg
- Mexico (7):
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Cuautla
  - Research Site, Guadalajara
  - Research Site, Guanajuato City
  - Research Site, Monterrey
  - Research Site, Veracruz
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Opole
  - Research Site, Oświęcim
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (9):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Galati
  - Research Site, Oradea
  - Research Site, Ploieşti
  - Research Site, Satu Mare
  - Research Site, Târgu Gânguleşti
  - Research Site, Timișoara
- Russia (3):
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Smolensk
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Helsingborg
  - Research Site, Rättvik
- Research Site, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Frias JP, Gonzalez-Galvez G, Johnsson E, Maaske J, Testa MA, Simonson DC, Dronamraju N, Garcia-Sanchez R, Peters AL. Efficacy and safety of dual add-on therapy with dapagliflozin plus saxagliptin versus glimepiride in patients with poorly controlled type 2 diabetes on a stable dose of metformin: Results from a 52-week, randomized, active-controlled trial. Diabetes Obes Metab. 2020 Jul;22(7):1083-1093. doi: 10.1111/dom.13997. Epub 2020 Mar 9. PMID 32052516
- See also: CV181365_CSP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4128&filename=CV181365_CSP.PDF

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 444 subjects were randomized in this international, multi-center study which was conducted at 88 centers in 10 countries between 14 Aug 2015 and 18 September 2019.
Pre-assignment Details: The study duration was up to 160 weeks, consisting of a 2-week screening period, 2-week lead-in period, 52-week short-term treatment period, and 104-week long-term treatment period (156-week treatment period). One subject did not start the short-term treatment period and so only 443 subjects received treatment.
Groups:
- Dapagliflozin 10mg and Saxagliptin 5mg: Subjects received dapagliflozin 10 mg, saxagliptin 5 mg plus placebo for glimepiride, each administered orally once daily. Subjects also continued to receive their metformin dose of at least 1500 mg per day
- Titrated Glimepiride: Subjects received titrated glimepiride 1, 2, 3, 4, or 6 mg plus placebo for saxagliptin and placebo for dapagliflozin, administered orally once daily. Subjects also continued to receive their metformin dose of at least 1500 mg per day.
Period: Short-term Treatment Period
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Started | 227 | 217
Recevied Treatment | 227 | 216
Completed | 210 | 194
Not Completed | 17 | 23
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Subject Request To Discontinue Treatment | 1 | 1
Not completed — Non-compliance with Study Drug | 0 | 2
Not completed — Worsening of liver function | 0 | 1
Not completed — Subject moved out of state | 0 | 1
Period: Long-term Treatment Period
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Started | 196 (Not all subjects who completed the previous period were eligible to enter the long-term period.) | 186 (Not all subjects who completed the previous period were eligible to enter the long-term period.)
Received Treatment | 196 | 183
Completed | 174 | 164
Not Completed | 22 | 22
Not completed — Non-compliance with Study Drug | 1 | 1
Not completed — Lost to Follow-up | 6 | 4
Not completed — Lack of Efficacy | 1 | 1
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 5
Not completed — Other | 4 | 4
Not completed — Subject Decision | 2 | 4
Not completed — Withdrawal by Subject | 8 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the randomized subjects data set which included all randomized subjects who received at least 1 dose of study medication during the double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride | Total
Number analyzed (Participants) | 227 | 216 | 443
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (10.11) | 56.1 (9.23) | 56.1 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 115 | 225
  Male | 117 | 101 | 218
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 11 | 10 | 21
  Black Or African American | 4 | 5 | 9
  Native Hawaiian Or Other Pacific Islander | 0 | 1 | 1
  Other | 6 | 4 | 10
  White | 206 | 196 | 402

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 52
Description: To examine whether the mean change from baseline in HbA1c with co-administered saxagliptin 5 mg and dapagliflozin 10 mg plus metformin is superior to titrated glimepiride plus metformin after 52 weeks of double-blind treatment.
Time Frame: Baseline and Week 52
Population: The randomized subject data set included all randomized subjects who received at least 1 dose of study medication during the double-blind treatment period. Of these, only subjects with an evaluable baseline measurement for a given endpoint were analysed.
Measure: Least Squares Mean (95% Confidence Interval); unit: % HbA1c
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Number analyzed (Participants) | 218 | 212
% HbA1c | -1.35 [-1.49 to -1.22] | -0.98 [-1.12 to -0.84]
Statistical Analysis 1: Comparison: Dapagliflozin 10mg and Saxagliptin 5mg vs Titrated Glimepiride; Test type: Superiority; p < 0.001, Mixed Models Analysis; Adjusted for for treatment, baseline HbA1c, visit, treatment-by-visit interaction, and baseline HbA1c-by-visit interaction; Least Squares (LS) Mean Difference = -0.37, 95% CI 2-sided [-0.57 to -0.18], Standard Error of Mean 0.099

2. Secondary Outcome: Change From Baseline in Total Body Weight at Week 52
Description: To examine whether the mean change from baseline in total body weight with co-administered saxagliptin 5 mg and dapagliflozin 10 mg plus metformin is superior to titrated glimepiride plus metformin after 52 weeks of double-blind treatment.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram (kg)
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Number analyzed (Participants) | 224 | 214
kilogram (kg) | -3.11 [-3.65 to -2.57] | 0.95 [0.38 to 1.51]
Statistical Analysis 1: Comparison: Dapagliflozin 10mg and Saxagliptin 5mg vs Titrated Glimepiride; Test type: Superiority; p < 0.001, Mixed Models Analysis; Adjusted for for treatment, baseline body weight, visit, treatment-by-visit interaction, and baseline body weight-by-visit interaction; LS Mean Difference = -4.06, 95% CI 2-sided [-4.84 to -3.28], Standard Error of Mean 0.397

3. Secondary Outcome: Percentage of Subjects Achieving a Therapeutic Glycemic Response, Defined as HbA1c < 7.0%, at Week 52
Description: Therapeutic glycemic response was defined as HbA1c <7.0%. Subjects rescued or discontinued prior to, and subjects with missing measurements at Week 52 were treated as non-responders. The percentage of subjects with a therapeutic glycemic response is based on the logistic regression method with adjustment for baseline HbA1c.
Time Frame: At Week 52
Population: The randomized subject data set included all randomized subjects who received at least 1 dose of study medication during the double-blind treatment period.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Number analyzed (Participants) | 227 | 216
Percentage of subjects | 44.3 [37.45 to 51.32] | 34.3 [27.87 to 41.33]
Statistical Analysis 1: Comparison: Dapagliflozin 10mg and Saxagliptin 5mg vs Titrated Glimepiride; Test type: Superiority; p = 0.044, Regression, Logistic; Adjusted for baseline HbA1c value; Odds Ratio (OR) = 1.5, 95% CI [1.01 to 2.29]

4. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 52
Description: To examine whether the change from baseline in SBP with co-administered saxagliptin 5 mg and dapagliflozin 10 mg plus metformin is superior to titrated glimepiride plus metformin after 52 weeks of double-blind treatment.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Number analyzed (Participants) | 224 | 214
mmHg | -2.6 [-4.4 to -0.8] | 1.0 [-0.9 to 2.9]
Statistical Analysis 1: Comparison: Dapagliflozin 10mg and Saxagliptin 5mg vs Titrated Glimepiride; Test type: Superiority; p = 0.007, Mixed Models Analysis; Adjusted for treatment, baseline SBP, visit, treatment-by-visit interaction, and baseline SBP-by-visit interaction; LS Mean Difference = -3.6, 95% CI 2-sided [-6.3 to -1.0], Standard Error of Mean 1.35

5. Secondary Outcome: Percentage of Subjects With Treatment Intensification During the 52-week Short-term Treatment Period
Description: Treatment intensification was defined as the addition of insulin or other glucose-lowering agent for rescue therapy or discontinuation for lack of glycemic control. Time to treatment intensification was censored after the 52-week treatment period if treatment intensification had not occurred by then. Subjects rescued at Week 52 were counted as having an event for the analysis. The values presented are the percentage of subjects requiring the addition of insulin or other glucose-lowering agent for rescue therapy or discontinuation for lack of glycemic control during the 52-week short -term treatment period.
Time Frame: Up to Week 52
Population: as for outcome 3
Measure: Number; unit: Percentage of Subjects
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Number analyzed (Participants) | 227 | 216
Percentage of Subjects | 1.3 | 8.8
Statistical Analysis 1: Comparison: Dapagliflozin 10mg and Saxagliptin 5mg vs Titrated Glimepiride; Time to treatment intensification was analyzed using a Cox proportional hazards model; Test type: Superiority; p = 0.002, Regression, Cox Proportional Hazards — This endpoint did not meet the required number of events (n=10) in each treatment arm, hence was excluded from sequential testing; Hazard Ratio (HR) = 0.15, 95% CI 2-sided [0.04 to 0.50]

6. Secondary Outcome: Percentage of Subjects With Treatment Intensification During the 156-Week Short-term Plus Long-Term Treatment Period.
Description: Treatment intensification was defined as the addition of insulin or other glucose-lowering agent for rescue therapy or discontinuation for lack of glycemic control. Time to treatment intensification was censored after 156-week treatment period if treatment intensification had not occurred by then. Subjects rescued at Week 156 were counted as having an event for the analysis. The values presented are the percentage of subjects requiring the addition of insulin or other glucose-lowering agent for rescue therapy or discontinuation for lack of glycemic control during the 156-week treatment period.
Time Frame: Up to Week 156
Population: as for outcome 3
Measure: Number; unit: Percentage of Subjects
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Number analyzed (Participants) | 227 | 216
Percentage of Subjects | 37.0 | 55.6
Statistical Analysis 1: Comparison: Dapagliflozin 10mg and Saxagliptin 5mg vs Titrated Glimepiride; Time to treatment intensification was analyzed using a Cox proportional hazards model; Test type: Superiority; p < 0.001, Regression, Cox Proportional Hazards; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.39 to 0.68]

7. Secondary Outcome: Percentage of Subjects Achieving a Therapeutic Glycemic Response, Defined as HbA1c < 7.0%, at Week 156
Description: Therapeutic glycemic response was defined as HbA1c <7.0%. Subjects rescued or discontinued prior to, and subjects with missing measurements at Week 156 were treated as non-responders. The percentage of subjects with a therapeutic glycemic response is based on the logistic regression method with adjustment for baseline HbA1c.
Time Frame: At Week 156
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Number analyzed (Participants) | 227 | 216
Percentage of Subjects | 21.4 [16.30 to 27.64] | 11.7 [8.03 to 16.82]
Statistical Analysis 1: Comparison: Dapagliflozin 10mg and Saxagliptin 5mg vs Titrated Glimepiride; Test type: Superiority; p = 0.006, Regression, Logistic; Adjusted for baseline HbA1c value; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.23 to 3.42], Standard Error of Mean 0.54

8. Secondary Outcome: Time to Treatment Intensification During the 156-Week Short-term Plus Long-Term Treatment Period.
Description: Treatment intensification was defined as the addition of insulin or other glucose-lowering agent for rescue therapy or discontinuation for lack of glycemic control. Time to treatment intensification was censored after 156-week treatment period if treatment intensification had not occurred by then. Subjects rescued at Week 156 were counted as having an event for the analysis. Time to treatment intensification curves were generated using Kaplan-Meier estimates and compared using a Cox proportional hazards model.
Time Frame: Up to Week 156
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
Number analyzed (Participants) | 227 | 216
Weeks | NA [NA to NA] — Not calculable as less than 50% of the subjects took rescue therapy or discontinued for lack of glycemic control before Week 156. | 92.3 [73.0 to 105.7]
Statistical Analysis 1: Comparison: Dapagliflozin 10mg and Saxagliptin 5mg vs Titrated Glimepiride; Test type: Superiority; p < 0.001, Regression, Cox Proportional Hazards; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.39 to 0.68]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs), including serious adverse events (SAEs), were collected on or after the date of first dose of short-term study medication and up to and including 4 days (other AEs) or 30 days (SAEs) after last dose. Up to a total of 160 weeks.
Description: The treated subjects data set for the short-tem plus long-term treatment period consisted of all subjects who received at least 1 dose of double-blind study medication during the short-term double-blind treatment period.
Arm/Group | Dapagliflozin 10mg and Saxagliptin 5mg | Titrated Glimepiride
All-Cause Mortality (participants affected / at risk) | 1/227 | 3/216
Serious Adverse Events (participants affected / at risk) | 29/227 | 24/216
Other Adverse Events (participants affected / at risk) | 99/227 | 106/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg and Saxagliptin 5mg (N=227) | Titrated Glimepiride (N=216)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (3) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (3)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Abdominal wall infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1)
Hormone level abnormal (Investigations) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg and Saxagliptin 5mg (N=227) | Titrated Glimepiride (N=216)
Upper respiratory tract infection (Infections and infestations) | 23 (29) | 21 (27)
Headache (Nervous system disorders) | 18 (21) | 16 (20)
Hypertension (Vascular disorders) | 7 (7) | 18 (18)
Bronchitis (Infections and infestations) | 11 (15) | 17 (21)
Influenza (Infections and infestations) | 9 (10) | 12 (16)
Nasopharyngitis (Infections and infestations) | 14 (20) | 19 (25)
Pharyngitis (Infections and infestations) | 6 (9) | 12 (13)
Urinary tract infection (Infections and infestations) | 31 (41) | 21 (28)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 13 (14)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 12 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (16) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT02419612/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT02419612/SAP_002.pdf